CLINICAL TRIAL: NCT00893737
Title: An Open-label Study to Evaluate "Completeness of Response" Following Treatment With Treximet™ for Migraine
Brief Title: "Completeness of Response" Following Treatment With Treximet™ for Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Roger K. Cady, MD, Clinvest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110211
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Migraine
Keywords: Migraine; Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treximet (Experimental): Treximet (a combination of sumatriptan 85 mg and naproxen sodium 500 mg) 1 tablet to be administered as soon as patient has headache indicative of migraine. Patient may treat up to 16 migraine attacks in 2 month study period.
  Interventions: Drug: sumatriptan succinate 85 mg/naproxen sodium 500 mg (Treximet)

INTERVENTIONS:
Drug: sumatriptan succinate 85 mg/naproxen sodium 500 mg (Treximet) — Treximet 1 tablet as soon as the patient has headache indicative of migraine. May be repeated between 2 and 24 hours post-treatment for persistent or recurring headache. Subjects should not take more than 2 Treximet tablets in 24 hours.

SUMMARY:
Many clinical trials may not fully explore criteria that are important to some migraine patients' definition of "complete response." This study offers the opportunity to evaluate the effectiveness of Treximet™ when non-standard criteria are examined (for example, neck pain, irritability or fatigue). Subjects enrolled at 8 investigative sites will complete 2 visits. Subjects will complete a Completeness of Response Survey at Visit 1 considering their usual migraine medication (a triptan) and a Completeness of Response Survey at Visit 2 considering their study medication (Treximet™).

DETAILED DESCRIPTION:
At the screening visit (Visit 1), following written informed consent, subjects will provide a medical, medication and migraine history. A physical and neurological exam and pregnancy test (if appropriate) will be performed. Vital signs will be recorded for all subjects. The Headache Impact Test (HIT-6) and Baseline Patient Perception of Migraine Questionnaire (PPMQ-R) will be completed with the Baseline Completeness of Response Survey (CORS) considering migraine therapy (triptan) utilized during the 3 months prior to enrollment. The Completeness of Response Survey will collect traditional and non-traditional symptoms. Subjects are instructed to treat all migraines that occur in the next 2 months. Subjects will treat with a single tablet of Treximet™ as soon as they have a headache indicative of migraine and are encouraged to treat when the headache is mild. A Headache Diary documenting onset of headache pain and associated symptoms, time of treatment with study medication, symptoms at 2 hours following treatment, time of relief, recurrence of symptoms within 24 hours post-treatment, and adverse events will be dispensed with study medication. Subjects may take a 2nd dose of study medication or medication determined by the investigator for rescue of persistent or recurring headache at 2 or more hours following the 1st dose of study medication. Alternate rescue medication can be provided at the discretion of the investigator but may not include triptan, non-steroidal anti-inflammatory (short-acting NSAID between 6 hours before and 2 hours after study medication or long-acting NSAID between 24 hours before and 24 hours after study medication), or ergotamine-containing or ergot-type medication. Subjects must be headache-free for 24 hours before recording the onset of a "new" migraine attack. The study coordinator will contact subjects at Month 1 to verify treatment and diary compliance.

At Visit 2, following 2 months of treatment with Treximet™, the subject will return to the study site and return completed Headache Diaries. The End of Study CORS, CORS Comparator and End of Study PPMQ-R will be completed considering response with study medication. Adverse events will be documented and Diaries and Questionnaires will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

Subject must be/have

* age 18 to 65
* able to read, understand, and sign informed consent
* willing to record migraine headaches and response to treatment in diary
* diagnosis of migraine headache (IHS 1.1 or 1.2), without and/or with aura
* at least one year history of migraine
* 3-8 attacks per month in past 3 months
* onset of migraine before age 50
* current triptan user (treated with triptan as primary migraine therapy at least 2 times per month in 3 months prior to screening)
* history of migraine starting at mild pain for at least 75% of migraine attacks
* use reliable method of birth control if female and childbearing potential (i.e. reliable barrier method, oral contraceptive, implant, contraceptive patch, long term injectable contraceptive, intrauterine device or tubal ligation)
* on stabilized dosages of current concomitant medications at least 90 days (may include migraine preventive medications), and willing to continue during study period

Exclusion Criteria:

Subject has/is

* history of serotonin syndrome
* medical condition that, in opinion of the investigator, could confound results of the study
* female of childbearing potential not using adequate contraceptive measures
* 15 or more headache days per month in total, or history of retinal,, basilar or hemiplegic migraine, cluster headache, or secondary headaches (such as due to trauma, infection, alterations of homeostasis, ENT or psychiatric disorders, cranial or cervical disorders or neuralgias)
* in investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or presence of risk factors including but not limited to, hypertension, hypercholesterolemia, smoker, obesity, diabetes, or family history of coronary artery disease)
* blood pressure ≥ 140/90 mmHg in 2 of 3 BP measurements at screening or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker
* a history of congenital heart disease, cardiac arrhythmias requiring medication, or history of clinically significant electrocardiogram abnormality that, in investigator's opinion, contraindicates participation in this study
* evidence or history of ischemic vascular disease including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with any of above
* evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower convulsive threshold; or has been treated with antiepileptic drug for seizure control within 5 years prior to screening
* history of impaired hepatic or renal function that, in investigator's opinion, contraindicates participation in study
* hypersensitivity, intolerance, or contraindication to use of any triptan, NSAID or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma
* currently taking, or has taken in previous three months, migraine prophylactic medication containing methysergide; or is taking migraine or menstrual migraine prophylactic medication that is not stabilized (i.e., change of dose within the past 2 months)
* recent history of regular use of opioids or barbiturates for treatment of migraine headache and/or other non-migraine pain (regular use defined as an average of 4 days per month over last 6 months)
* taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within 2 weeks prior to screening through 2 weeks post final study treatment
* history of any bleeding disorder or is currently taking anti-coagulant or antiplatelet agent
* evidence or history of gastrointestinal surgery or GI ulceration or perforation in past six months, gastrointestinal bleeding in past year; or evidence or history of inflammatory bowel disease
* pregnant, actively trying to become pregnant, or breast feeding
* evidence of alcohol or substance abuse within last year or any concurrent medical or psychiatric condition which, in investigator's judgment, will likely interfere with study conduct, subject cooperation, or evaluation and interpretation of study results, or which otherwise contraindicates participation in this clinical trial
* participated in an investigational drug trial within previous four weeks or plans to participate in another study at any time during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (8):
- United States (8):
  - San Francisco Clinical Research Center, San Francisco, California
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Clinvest, Springfield, Missouri
  - Mercy Health Research/Ryan Headache Center, St Louis, Missouri
  - Island Neurological Associates, PC, Plainview, New York
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Wesley Headache Clinic and Research Center, Cordova, Tennessee
  - Texas Headache Associates, San Antonio, Texas

REFERENCES:
- [Background] Smith TR, Sunshine A, Stark SR, Littlefield DE, Spruill SE, Alexander WJ. Sumatriptan and naproxen sodium for the acute treatment of migraine. Headache. 2005 Sep;45(8):983-91. doi: 10.1111/j.1526-4610.2005.05178.x. PMID 16109111
- [Background] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970
- [Background] Silberstein SD. Practice parameter: evidence-based guidelines for migraine headache (an evidence-based review) [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2000 Sep 26;55(6):754-62. doi: 10.1212/wnl.55.6.754. No abstract available. PMID 10993991
- [Derived] Cady R, Banks J, Nett RB, Goldstein J, Bennett N, Turner IM, Ruoff GE, Landy SH, Farmer K, Juhasz M, Tarrasch J, Runken MC. Multi-center comparison of response to a single tablet of sumatriptan 85 mg and naproxen 500 mg vs usual therapy treating multiple migraine attacks as measured by the completeness of response survey. Headache. 2011 Jun;51(6):961-70. doi: 10.1111/j.1526-4610.2011.01912.x. Epub 2011 May 17. PMID 21592098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In 6/2/09 Last Patient In 7/17/09 Patients enrolled at 5 Headache Specialty clinics, 2 Primary Care practices, and 1 Neurological practice.
Period: Overall Study
Arm/Group | Treximet
Started | 147
Completed | 135
Not Completed | 12
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treximet
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 145
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Secondary Outcome: Percent of Participants Reporting Treximet Provides Therapeutic Advantage Over Usual Pre-study Triptan
Description: CORS completed at Visit 1 regarding participant pre-study triptan and at Visit 2 regarding Treximet taken in study. Areas of therapeutic advantage evaluated: How often does 1 dose completely relieve (1) headache pain (2) neck/shoulder pain (3) nausea (4) light sensitivity (5) sound sensitivity (6) irritability. How quickly can/do you (1) concentrate or think clearly (2) resume normal activities (3) function normally (4) feel completely normal. How confident are you that (1) one dose will completely relieve migraine within 2 hours (2) once relieved, migraine will not return within 24 hours.
Time Frame: Visit 1 (screening) and Visit 2 (study completion following 2-month treatment period)
Measure: Number; unit: Percent of Participants
Arm/Group | Treximet
Number analyzed (Participants) | 147
Percent of Participants
  How often 1 dose relieves headache pain | 42
  How often 1 dose relieves neck/shoulder pain | 52
  How often 1 dose relieves nausea | 43
  How often 1 dose relieves light sensitivity | 42
  How often 1 dose relieves sound sensitivity | 45
  How often 1 dose relieves irritability | 36
  How quickly can you concentrate or think clearly | 31
  How quickly can you resume normal activities | 32
  How quickly can you function normally | 32
  How quickly do you feel completely normal | 36
  Confidence 1 dose will relieve migraine in 2 hours | 33
  Confidence migraine will not return in 24 hours | 38

2. Secondary Outcome: Paired T-test Indicating Greater Subject Satisfaction With Treximet Over Usual Pre-study Triptan as Determined by the Revised Patient Perception of Migraine Questionnaire (PPMQ-R)
Description: Scores calculated for (1) Efficacy (2) Functionality (3) Ease of use (4) Cost. Higher score represents better treatment satisfaction.
Time Frame: Visit 1 (screening) and Visit 2 (study completion following 2-month treatment period)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Treximet
Number analyzed (Participants) | 147
Units on a scale
  Efficacy | 8.61 [4.64 to 12.58]
  Functionality | 13.86 [9.39 to 18.32]
  Ease of Use | 2.76 [-0.11 to 5.64]
  Cost | 7.28 [1.83 to 12.72]

3. Primary Outcome: Change in Scores From Completeness of Response Survey (CORS)
Description: CORS scores for Pain (0-4), Associated Symptoms (0-4), Limbic/Affective Symptoms (0-5), and Speed of Return to Functionality (1-5), represent outcome measures that are relevant to patients. Higher scores represent better treatment efficacy.
  The analysis compares CORS scores for usual triptan (pre-study) versus (vs.) Treximet (study medication).
Time Frame: Visit 1 (screening) and Visit 2 (study completion following 2-month treatment period)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Treximet
Number analyzed (Participants) | 147
Units on a scale
  Pain Score | 0.17 [0.03 to 0.30]
  Associated Symptoms Score | 0.07 [-0.09 to 0.24]
  Limbic Symptoms Score | 0.03 [-0.12 to 0.18]
  Functionality Score | 0.10 [-0.05 to 0.26]

ADVERSE EVENTS:
Arm/Group | Treximet
Serious Adverse Events (participants affected / at risk) | 2/147
Other Adverse Events (participants affected / at risk) | 28/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treximet (N=147)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Migraine without aura (Nervous system disorders) | 1 (1) — without intractable headache, but with Status Migrainosus
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treximet (N=147)
Chest Tightness (General disorders) | 4 (8)
Dizziness (Nervous system disorders) | 5 (9)
Jittery (General disorders) | 3 (19)
Light Headed (Nervous system disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 9 (20)
Sleepy (Nervous system disorders) | 5 (21)
Tired (Nervous system disorders) | 4 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of Results is specifically authorized, subject to the provisions of STUDY AGREEMENT. INVESTIGATOR is free to publish Results of its part of study in collaboration with other investigators, but in compliance with confidentiality agreement and subsequent to full study publication issued by CLINVEST. INVESTIGATOR agrees to submit a copy of any results communication to CLINVEST for review and comment 60 days prior to submission for publication.